CLINICAL TRIAL: NCT02312596
Title: A Prospective, Randomized Clinical Trial of PRP Concepts Fibrin Bio-Matrix in Non-Healing Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PRP Concepts, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC002
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Foot Ulcers
Keywords: non-healing wound; diabetic foot ulcer; platelet rich plasma
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PRP Concepts Fibrin Bio-Matrix (Experimental): PRP Concepts Fibrin Bio-Matrix
  Interventions: Device: PRP Concepts Fibrin Bio-Matrix; Other: Usual and Customary Practice
- Usual and customary practice (Active Comparator): Usual and customary practice
  Interventions: Other: Usual and Customary Practice

INTERVENTIONS:
Device: PRP Concepts Fibrin Bio-Matrix — Application of PRP Concepts Fibrin Bio-Matrix in addition to usual and customary practice
  Arms: PRP Concepts Fibrin Bio-Matrix
Other: Usual and Customary Practice — Usual and customary care for non-healing wounds
  Other Names: Standard of Care

SUMMARY:
A prospective, randomized, controlled, clinical study to establish clinical based evidence of PRP Concepts Fibrin Bio-Matrix and compare its performance with the usual and customary practice for the treatment of Wagner 1 or 2 DFUs.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, controlled, multi-center study for subjects undergoing DFU treatment. Qualified subjects will be randomized (1:1); test group (PRP Concepts Fibrin Bio-Matrix) and control group (usual and customary practice). The study will consist of 3 periods: a screening period, an active treatment period, and a follow-up period (if healed). Approximately 250 subjects will be enrolled. Subjects will be ≥18 years of age with a chronic Wagner grade 1 or 2 DFU (greater than 1 month duration). Each subject will be enrolled in the active treatment period for up to 12 weeks, or to closure of wound with a confirmatory visit 2 weeks after wound closure, whether such closure occurs at 12 weeks or earlier.

ELIGIBILITY:
Inclusion Criteria:

* Medicare eligible
* A full thickness diabetic foot ulcer with a viable wound bed
* Diabetes mellitus (type I or II) that is adequately controlled
* The ulcer is greater than 4 weeks duration.
* The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (index ulcer) is a Wagner 1 or 2 DFU (see Appendix for Wagner Classification) that is located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces but not on the heel).
* Post-debridement, the ulcer size must be between 0.5 - 20 cm2.
* One of the following assessments was completed to confirm pedal circulation: ankle / brachial index is between 0.7 to 1.2; transcutaneous partial pressure oxygen (TcPO2) > 30 mmHg at the ankle; or toe pressure of >40mm Hg or a doppler waveform consistent with adequate flow in the foot (biphasic or triphasic)
* Able and willing to provide a voluntary written informed consent.
* Able and willing to wear an off-loading device or orthopedic shoe
* Able and willing to attend scheduled follow-up visits and study related exams

Exclusion Criteria:

* Greater than 30% reduction in wound size during the first two weeks of observation and treatment by the investigator
* Wagner 3, 4, 5 DFU
* Gross clinical infection at the study ulcer site including cellulitis and osteomyelitis
* Wounds that are likely to require dressing changes more frequent than twice weekly (heavy exudates).
* Known allergy tor sensitivity to Eclipse PRP kit components (calcium chloride, calcium gluconate or acid citrate dextrose solution A (ACDA))
* Presence of Gangrene
* Active Charcot's disease as determined by clinical and radiographic examination of a non-diabetic pathophysiology (e.g., rheumatoid, radiation-related, and vasculitis related ulcers)
* Malignancy at or near the ulcer site
* Known serum albumin < 2.5 mg/dl, Known renal failure as determined by a Creatinine > 2.5 mg/dl, Plasma Platelet count of less than 100 x 109/L, Hemoglobin of less than 10.5 g/dL
* Rheumatoid arthritis (and other collagen vascular disease), vasculitis, sickle cell disease, HIV
* Severe liver disease. Severe liver disease is defined as known history of chronic hepatitis or cirrhosis &/or the following abnormal Liver Function Tests: ALT & AST >35, ALP >120, PT >12 seconds.
* Presence of additional abnormal lab values obtained within 7 days prior to the Day 0 visit determined to be clinically significant by the investigator including: WBC >13,000/cm3 or < 5, 000 cm3, or electrolytes that are outside the host institution's range of normal.
* Radiation therapy, chemotherapy, chronic steroid use or immunosuppressive therapy within 30 days of enrollment
* Received another investigational device or drug within 30 days of enrollment
* Received allograft, autograft or xenograft within 30 days of enrollment
* Subject has inadequate venous access for repeated blood draw required for Eclipse RPR administrations
* Subject requires or is anticipated to require interventions directed at improvement of arterial perfusion to affected area.
* Ulcer expected to be treated with any advanced therapeutics (e.g., HBOT)
* Any condition judged by the investigator that would cause the study to be detrimental to the subject
* Alcohol or drug abuse, defined as current medical treatment for substance abuse
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound closure | 12 weeks
  Complete wound closure is defined as full epithelialization of the wound with the absence of drainage, durability confirmed at 2 weeks
Percent of wounds healed | 12 weeks
  Percentage of closure of the wound

SECONDARY OUTCOMES:
Wound Trajectory | 4, 8, 12 weeks
  Mean of percent (%) wound size changes at 4 weeks, 8 weeks and 12 weeks
Ulcer Recurrence | 3 months
  Ulcer recurrence out to 3 months for subjects whose wounds heal by conclusion of 12 week visit.
Quality of Life score | 3 months
  Changes in Quality of Life scores and ability to return to previous function/resumption of normal activities

CONTACTS AND LOCATIONS:
Overall Officials: Damon Keeley, Study Director — PRP Concepts, LLC
Locations (1):
- Westchester General Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No